CLINICAL TRIAL: NCT00045630
Title: A Sequential Approach to the Treatment of Muscle Invasive, Non-Metastatic Urothelial Carcinoma of the Bladder: A Phase II Trial of Neoadjuvant Gemcitabine, Paclitaxel and Carboplatin With Molecular Correlates
Brief Title: S0219, Combination Chemotherapy Followed By Observation or Surgery in Patients With Stage II or Stage III Cancer of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256921; S0219 (Other: SWOG); U10CA032102 (NIH); NCT00191217 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-04

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: anterior urethral cancer; localized transitional cell cancer of the renal pelvis and ureter; posterior urethral cancer; stage II bladder cancer; stage III bladder cancer; transitional cell carcinoma of the bladder; urethral cancer associated with invasive bladder cancer; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Carboplatin; Gemcitabine; Paclitaxel; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine, Paclitaxel, Carboplatin (Experimental): Gemcitabine, Paclitaxel, Carboplatin followed by surgery
  Interventions: Drug: carboplatin; Drug: gemcitabine; Drug: paclitaxel; Procedure: surgery

INTERVENTIONS:
Drug: carboplatin
Drug: gemcitabine
  Other Names: gemcitabine hydrochloride
Drug: paclitaxel
  Other Names: Taxol
Procedure: surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells and decrease the need for surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by observation or surgery to remove the bladder (cystectomy) in treating patients who have stage II or stage III cancer of the urothelium.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the pathologic complete response of patients with stage II or III transitional cell cancer of the urothelium treated with neoadjuvant gemcitabine, paclitaxel, and carboplatin followed by observation or immediate cystectomy.
* Determine, preliminarily, if molecular markers predict response, survival, and tumor recurrence in patients treated with these regimens.
* Determine recurrence rates and cystectomy-free survival of patients who choose observation after an initial response to neoadjuvant chemotherapy.
* Compare the survival of patients treated with neoadjuvant chemotherapy followed by cystectomy vs observation.
* Determine the feasibility, tolerability, and toxicity of these regimens in these patients.

OUTLINE: This is a multicenter study.

Patients receive gemcitabine IV over 30 minutes and paclitaxel IV over 30 minutes on days 1 and 8 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Within 4-8 weeks after completion of neoadjuvant chemotherapy, patients undergo a third transurethral resection of bladder tumor.

Patients with T0 disease after neoadjuvant chemotherapy may choose to undergo observation. These patients undergo cystoscopies with biopsies every 3 months for 1 year, every 4 months for 1 year, and then every 6 months until disease progression.

Patients with T1 disease or greater after neoadjuvant chemotherapy undergo immediate cystectomy. Patients with T0 disease may also choose this option. Patients undergoing immediate cystectomy are followed every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 95 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed muscle-invasive (T2-T4a), node-negative (N0) urothelial transitional cell cancer (TCC) of the bladder
* Focal squamous and/or adenocarcinoma differentiation, defined as ≤ 10% of tumor volume allowed
* The following diagnoses are not allowed:

  * Small cell carcinoma
  * Sarcomatoid components
* Disease diagnosed with an initial transurethral resection of bladder tumor (TURBT) and a second TURBT performed within 8 weeks of first with attempt to remove all tumor present

  * Residual disease after second TURBT allowed
  * No more than 14-56 days after second TURBT
* No metastatic disease by chest x-ray and CT scan or MRI of the abdomen and pelvis
* Fresh tumor tissue, paraffin tumor tissue, unstained slides, or cell block specimen from one or both TURBTs available

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* White blood cell count (WBC) at least 3,500/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least lower limit of normal

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* Aspartate aminotransferase (SGOT) no greater than 2 times upper limit of normal

Renal

* Creatinine no greater than 2.0 mg/dL AND/OR
* Creatinine clearance at least 60 mL/min

Other

* No prohibitive medical risk that would preclude radical cystectomy
* No other serious concurrent systemic disorder that would preclude study compliance
* No other malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer in complete remission, or any other cancer for which patient has been disease-free for 5 years
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Prior intravesical immunotherapy allowed

Chemotherapy

* No prior systemic chemotherapy for TCC of the urothelium
* Prior intravesical chemotherapy allowed

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for TCC of the urothelium
* No concurrent radiotherapy

Surgery

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-01; Primary Completion 2008-05 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Primo N. Lara, MD, Study Chair — University of California, Davis
Locations (128):
- United States (128):
  - Cancer Center at Providence Alaska Medical Center, Anchorage, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Desert Medical Center, Mesa, Arizona
  - Banner Baywood Medical Center, Mesa, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Cancer Center at Vail Valley Medical Center, Edwards, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Forsyth Regional Cancer Center at Forsyth Medical Center, Winston-Salem, North Carolina
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - AnMed Health Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - University of Tennessee Cancer Institute - Medical Center, Memphis, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] deVere White RW, Lara PN Jr, Goldman B, Tangen CM, Smith DC, Wood DP Jr, Hussain MH, Crawford ED. A sequential treatment approach to myoinvasive urothelial cancer: a phase II Southwest Oncology Group trial (S0219). J Urol. 2009 Jun;181(6):2476-80; discussion 2480-1. doi: 10.1016/j.juro.2009.01.115. Epub 2009 Apr 16. PMID 19371909
- [Result] Lara PN, Goldman B, De Vere White R, et al.: A sequential treatment approach to muscle-invasive urothelial cancer: A phase II Southwest Oncology Group trial (S0219) of neoadjuvant paclitaxel, carboplatin, and gemcitabine (PCG). [Abstract] J Clin Oncol 26 (Suppl 15): A-5022, 2008.

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery: Patients receive 3 cycles (1 cycle = 21 days) of neoadjuvant chemotherapy (800 mg/m^2 of gemcitabine IV and 80 mg/m^2 of Paclitaxel IV on days 1 and 8 and Carboplatin IV on day 1), TURBT within 4-8 weeks of chemotherapy, option of proceeding with immediate cystectomy or observation.
Period: Overall Study
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Started | 77
Eligible | 75
Eligible and Began Protocol Therapy | 74
Completed | 71
Not Completed | 6
Not completed — Adverse Event | 1
Not completed — Refusal unrelated to adverse event | 1
Not completed — Progression/relapse | 1
Not completed — Death | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Number analyzed (Participants) | 74
Age Continuous [Median (Full Range); unit: years] | 69 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 55
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 70
  More than one race | 0
  Unknown or Not Reported | 0
Performance Status [Number; unit: participants] — Patients will be graded according to the Zubrod performance status scale. 0: Fully active, able to carry all pre-disease performance without restriction. 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. 2: Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours. 3: Capable of limited self-care, confined to bed or chair more than 50% of waking hours. 4: Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  participants
    0 | 50
    1 | 16
    Missing | 8
Clinical T Stage [Number; unit: participants] — Primary Tumor (T): TX Primary tumor cannot be assessed, T0 No evidence of primary tumor, Ta Non-invasive papillary carcinoma, Tis Carcinoma in situ: "flat tumor", T1 Tumor invades subepithelial connective tissue, T2 Tumor invades muscle, pT2a Tumor invades superficial muscle (inner half), pT2b Tumor invades deep muscle (outer half), T3 Tumor invades perivesical tissue, pT3a Microscopically, pT3b Macroscopically (extravesical mass), T4 Tumor invades any of the following: prostate, uterus, vagina, pelvic wall, abdominal wall, T4a Tumor invades prostate, uterus, vagina.
  participants
    T2 | 52
    T3 | 17
    T4a | 5
Prior Intravesical Therapy [Number; unit: participants]
  Yes | 11
  No | 59
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate by Transurethral Resection of Bladder Tumor (TURBT) and Imaging Studies After Chemotherapy
Description: Pathologic complete response (CR) is defined as absence of viable tumor in the TURBT specimen. Stable/No Response is defined as at least some disease evaluation tests were done (same tests as baseline) and status does not qualify for CR or Progression. Progression is defined as one or more of the following must occur: unequivocal progression of disease in the opinion of the treating physician. Appearance of any new lesion/site. Death due to disease without documented progression or symptomatic deterioration.
Time Frame: up to 12 weeks after registration (assessed within 8 weeks after completion of 3 cycles of chemotherapy )
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Number analyzed (Participants) | 74
percentage of participants | 46 [34 to 58]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined from the date of registration to date of death from any cause
Time Frame: 0-2 years
Population: All eligible patients who started treatment were included in the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Number analyzed (Participants) | 74
percentage of participants | 59 [45 to 72]

3. Secondary Outcome: Number of Patients With Grade 3 Through Grade 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 2.0. For each patient, worst grade of each event type is reported. Grade 3 = Severe, Grade 4 = Life-threatening, Grade 5 = Fatal.
Time Frame: Patients were assessed for adverse events at weeks 1, 2, 4, 5, 7, 8, and following surgery
Population: Eligible patients who had received any treatment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Number analyzed (Participants) | 74
Participants
  Abnormal troponin I (cTnI) | 1
  Allergic reaction | 2
  Anemia | 5
  Bilirubin increase | 1
  Cardiac ischemia/infarction | 1
  Creatinine increase | 1
  Diarrhea without colostomy | 2
  Duodenal ulcer | 1
  Dyspnea | 1
  Fatigue/malaise/lethargy | 3
  Febrile neutropenia | 2
  GI-other | 1
  Hemolysis | 1
  Incontinence | 1
  Infection with 3-4 neutropenia | 2
  Infection, unk ANC | 2
  Leukopenia | 22
  Lymphopenia | 1
  Melena/ GI bleeding | 1
  Neutropenia/granulocytopenia | 41
  SGPT (ALT) increase | 1
  Thrombocytopenia | 13
  Ureteral obstruction | 1
  Urinary tr infect w/ neutrop | 1
  Urinary tr infect w/o neutrop | 1
  Vomiting | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events at weeks 1, 2, 4, 5, 7, 8, and following surgery
Arm/Group | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery
Serious Adverse Events (participants affected / at risk) | 2/74
Other Adverse Events (participants affected / at risk) | 73/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery (N=74)
GI-other (Gastrointestinal disorders) | 1
Infection with 3-4 neutropenia (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine, Paclitaxel, Carboplatin Followed by Surgery (N=74)
Anemia (Blood and lymphatic system disorders) | 49
Blurred vision (Eye disorders) | 5
Abdominal pain/cramping (Gastrointestinal disorders) | 8
Constipation/bowel obstruction (Gastrointestinal disorders) | 21
Diarrhea without colostomy (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 31
Stomatitis/pharyngitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 9
Edema (General disorders) | 7
Fatigue/malaise/lethargy (General disorders) | 61
Fever without neutropenia (General disorders) | 8
Pain-other (General disorders) | 14
Rigors/chills (General disorders) | 9
Allergic reaction (Immune system disorders) | 6
Infection w/o 3-4 neutropenia (Infections and infestations) | 6
Infection, unk ANC (Infections and infestations) | 4
Urinary tr infect w/o neutrop (Infections and infestations) | 6
Creatinine increase (Investigations) | 7
Leukopenia (Investigations) | 48
Lymphopenia (Investigations) | 6
Neutropenia/granulocytopenia (Investigations) | 54
SGOT (AST) increase (Investigations) | 11
SGPT (ALT) increase (Investigations) | 15
Thrombocytopenia (Investigations) | 41
Weight loss (Investigations) | 8
Anorexia (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dizziness/light headedness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Sensory neuropathy (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 4
Dysuria (Renal and urinary disorders) | 4
Hematuria (Renal and urinary disorders) | 4
Urinary frequency/urgency (Renal and urinary disorders) | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 36
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No